CLINICAL TRIAL: NCT01110616
Title: A Double Blind, Randomized, Crossover Study to Assess EEG Platform Standardization in Healthy Male Subjects
Brief Title: EEG (Electroencephalogram) Platform Standardization in Healthy Male Subjects (3134-010)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3134-010; MK3134-010
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Dementia
Keywords: EEG Standardization
MeSH Terms: conditions — Dementia | interventions — Lorazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- Sequence 1 (Experimental): MK3134-Lorazepam-Placebo-MK3134-Lorazepam
  Interventions: Drug: MK3134; Drug: Comparator: Lorazepam; Drug: Comparator: Placebo
- Sequence 2 (Experimental): MK3134-Lorazepam-Placebo-Lorazepam-MK3134
  Interventions: Drug: MK3134; Drug: Comparator: Lorazepam; Drug: Comparator: Placebo
- Sequence 3 (Experimental): MK3134-Placebo-Lorazepam-MK3134-Lorazepam
  Interventions: Drug: MK3134; Drug: Comparator: Lorazepam; Drug: Comparator: Placebo
- Sequence 4 (Experimental): MK3134-Placebo-Lorazepam-Lorazepam-MK3134
  Interventions: Drug: MK3134; Drug: Comparator: Lorazepam; Drug: Comparator: Placebo
- Sequence 5 (Experimental): Lorazepam-Placebo-MK3134-MK3134-Lorazepam
  Interventions: Drug: MK3134; Drug: Comparator: Lorazepam; Drug: Comparator: Placebo
- Sequence 6 (Experimental): Lorazepam-Placebo-MK3134-Lorazepam-MK3134
  Interventions: Drug: MK3134; Drug: Comparator: Lorazepam; Drug: Comparator: Placebo
- Sequence 7 (Experimental): Lorazepam-MK3134-Placebo-MK3134-Lorazepam
  Interventions: Drug: MK3134; Drug: Comparator: Lorazepam; Drug: Comparator: Placebo
- Sequence 8 (Experimental): Lorazepam-MK3134-Placebo-Lorazepam-MK3134
  Interventions: Drug: MK3134; Drug: Comparator: Lorazepam; Drug: Comparator: Placebo
- Sequence 9 (Experimental): Placebo-MK3134-Lorazepam-MK3134-Lorazepam
  Interventions: Drug: MK3134; Drug: Comparator: Lorazepam; Drug: Comparator: Placebo
- Sequence 10 (Experimental): Placebo-MK3134-Lorazepam-Lorazepam-MK3134
  Interventions: Drug: MK3134; Drug: Comparator: Lorazepam; Drug: Comparator: Placebo
- Sequence 11 (Experimental): Placebo-Lorazepam-MK3134-MK3134-Lorazepam
  Interventions: Drug: MK3134; Drug: Comparator: Lorazepam; Drug: Comparator: Placebo
- Sequence 12 (Experimental): Placebo-Lorazepam-MK3134-Lorazepam-MK3134
  Interventions: Drug: MK3134; Drug: Comparator: Lorazepam; Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK3134 — MK3134, 25 mg tablets (5 x 5 mg capsule), orally
Drug: Comparator: Lorazepam — Lorazepam, 2 mg (2 x 1 mg tablet), orally
  Other Names: Lorazepam
Drug: Comparator: Placebo — Placebo, to match MK3134, and placebo to match Lorazepam

SUMMARY:
The objective of this study is to test the experimental reproducibility and within-subject variability of qEEG (quantitative electroencephalogram) using two probe compounds: MK3134 and lorazepam.

This study will test the hypothesis that EEG (Electroencephalogram) theta power, averaged across a topographical region of interest is decreased 6 hours after administration of MK3134 compared to placebo.

The objective of this study is to test the experimental reproducibility and within-subject variability of qEEG using two probe compounds: MK3134 and lorazepam.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male between 18 to 40 years of age
* The subject has a Body Mass Index (BMI) greater than or equal to 31 kg/m^2 at the prestudy (screening) visit
* Subject has normal or corrected to normal visual and auditory acuity
* Subject has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months
* Subject is right-handed

Exclusion Criteria:

* Subject has permanent cosmetic or metallic objects in their body that can interfere with the measurements
* Subject has a history of stroke, chronic seizures, or major neurological disorder
* Subject has a history of neoplastic disease
* Subject has a current diagnosis of or a prior history of sleep apnea
* Subject has a history of fainting during blood draws
* Subject has a history of significant head injury/trauma
* Subject has a current diagnosis of or history of Bipolar illness, Schizophrenia, Attention Deficit Hyperactivity Disorder (ADHD), or claustrophobia
* Subject works a night shift and is not able to avoid night shift work within 3 days before each treatment visit
* Subject is currently a regular user of any illicit drugs or has a significant history of drug (including alcohol) abuse

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
EEG (Electroencephalogram) theta power averaged across a topographical region of interest 6 hours after administration of MK3134/placebo | Baseline and 6 hours

SECONDARY OUTCOMES:
EEG (Electroencephalogram) beta and sigma power averaged across all cortical leads 2 hours after administration of lorazepam/placebo | Baseline and 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC